CLINICAL TRIAL: NCT02265198
Title: Relationship of Pulmonary Contusion Morphology to Pulmonary Inflammation and Incidence of Acute Respiratory Distress Syndrome
Brief Title: Relationship of Pulmonary Contusion to Pulmonary Inflammation and Incidence of Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: BG03-018
Record Dates: First submitted 2014-10-07; First posted 2014-10-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-10

CONDITIONS: Pulmonary Contusion; Respiratory Failure; ARDS
Keywords: Pulmonary Contusion; ARDS; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchial Alveolar Lavage - Supernatant Blood-Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- PC Group: patients with Pulmonary Contusion on chest computed tomography (CT)
- Control Group 1: Uninjured patients undergoing elective surgical procedures that will require intubation and mechanical ventilation
- Control Group 2: Trauma patients without chest injury who are mechanically ventilated
- MICU group: Patients in the Medical ICU who are mechanically ventilated with acute respiratory failure

SUMMARY:
Pulmonary contusion (PC) is a significant problem after blunt trauma that may often lead to acute respiratory distress syndrome (ARDS) and in some patients, death. Although the pathophysiology is incompletely understood, it is clear that there is a biochemical process involving changes in the inflammatory milieu after contusion which occurs in addition to simple direct mechanical injury to the lung. The relationship of severity of contusion on imaging, disturbances in the inflammatory phenotype, and outcome is unknown. This is a prospective, observational study which will evaluate the size and severity of contusion as measured on chest computed tomography (CT). Inflammatory mediators will be measured in the bronchoalveolar lavage (BAL) and in the serum of patients with pulmonary contusion to define the inflammatory nature of the post-contusion lung. The degree of abnormality within the inflammatory parameters will be correlated with lung contusion size and subsequent patient outcomes. These data will be compared to other patient groups: 1) Trauma patients without chest injury who are mechanically ventilated; 2) Uninjured patients undergoing elective surgical procedures that will require intubation and mechanical ventilation; 3) Patients in the Medical ICU who are mechanically ventilated with acute respiratory failure.

The hypothesis tested within this study is resolution of lung injury is dependent upon the presence of Tregs in the alveolar space.

DETAILED DESCRIPTION:
The study will be conducted at Wake Forest University Baptist Medical Center and will enroll 40 patients in the PC study group, 20 patients in each control group, and 20 MICU patients. Recruitment will occur over two years. The sample size was determined by identifying the mean number of patients with PC admitted (38) to WFUBMC per year. Using Whittemore's formula, this sample size will be adequate to detect a significant odds ratio of 5 (alpha <0.05) with respect to increase in acute lung injury or ARDS risk in patients with > 20 % total lung volume contusion with approximately 85% power. The odds ratio for this population in developing acute lung injury or ARDS in a previous study was 16.666. Eligible subjects for study group will be patients with PC on admission CT; eligible subjects for control group #1 (CG1) are non-injured patients without PC undergoing a standard general surgical procedure; eligible subjects for control group #2 (CG2) are non-chest, non-PC trauma patients who are admitted intubated to the trauma ICU; eligible MICU subjects are patients on mechanical ventilation admitted to the Medical ICU with acute respiratory failure.

Informed consent for study group, CG2, and the MICU group will generally be obtained from family members as most patients will be unconscious or sedated. If the patient is alert, the study will be explained to both the patient and family. Informed consent for CG1 will be obtained from the patient and family members in Surgery Clinic prior to elective procedures. An initial blood sample will be obtained on all persons in the study group, CG2, and, if the patient is ventilated, a BAL will be obtained after signing of the informed consent by the patient or LAR. Blood samples and pulmonary samples will be obtained on CG1 patients after obtaining signed informed consent, in the operating theater, after they are sedated and intubated, though before their elective procedure. Blood and pulmonary samples will be obtained from MICU subjects after obtaining signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age > 15 years old
* Chest trauma patients
* Medical ICU patients with respiratory failure
* Elective surgery patients
* Trauma or surgical ICU patients on ventilators without chest trauma/pulmonary contusion

Exclusion Criteria:

* Age 15 years and younger
* Pregnant women
* Subjects with multiple myeloma, pheochromocytoma, homozygous sickle cell disease, or thyroid disorders
* Traumatic brain injury requiring intracranial pressure monitoring
* Moribund status

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at Wake Forest University Baptist Medical Center and will enroll 40 patients in the PC study group, 20 patients in each control group, and 20 MICU patients. Eligible subjects for study group will be patients with PC on admission CT; eligible subjects for control group #1 (CG1) are normal patients without PC undergoing a standard general surgical procedure; eligible subjects for control group #2 (CG2) are non-chest, non-PC trauma patients who are admitted intubated to the trauma ICU; eligible MICU subjects are patients on mechanical ventilation admitted to the Medical ICU with acute respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Volume of Pulmonary Contusion on CT scan | 14 days
  Measured volume of pulmonary contusion on CT scan correlates with increase in ventilator free days, ICU days, hospital days, and mortality
Volume of serum inflammatory mediator levels in BAL fluid | 14 days
  Volume of serum inflammatory mediator levels correlates with increase in ventilator free days, ICU days, hospital days, and mortality

SECONDARY OUTCOMES:
Presence of Tregs in BAL fluid | 14 days
  Measure presence of Tregs in BAL (% or absolute) to determine if positively correlated with reduced lung injury duration (increase in ventilator free days)
Presence of activated neutrophils in BAL fluid | 14 day
  measure neutrophil phenotypes in numbers to determine correlation with vent free days and mortality
Appearance of M2 macrophage phenotypes in BAL fluid | 14 day
  measure macrophage phenotype (M1 or M2) numbers and percent to determine correlation with vent free days and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hoth, MD, Principal Investigator — Wake Forest University Health Sciences; Peter E Morris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No